CLINICAL TRIAL: NCT00002407
Title: A Randomized Open-Label Strategic Study to Evaluate the Safety and Efficacy of 3 Different Convergent and Divergent Drug Combination Therapies in Anti-Retroviral Naive HIV-1 Infected Patients With CD4+ Counts Above 200/mm3
Brief Title: A Study of Three Drug Combination Therapies in HIV-Infected Patients Who Have Never Been Treated With Anti-HIV Drugs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: ATLANTIC STUDY
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1998-11

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Indinavir; Nevirapine; Lamivudine; Stavudine; Didanosine

INTERVENTIONS:
Drug: Indinavir sulfate
Drug: Nevirapine
Drug: Lamivudine
Drug: Stavudine
Drug: Didanosine

SUMMARY:
The purpose of this study is to see if it is safe and effective to give one of three different triple-drug combinations to HIV-infected patients who have never been treated with anti-HIV drugs.

DETAILED DESCRIPTION:
In this open-label, strategic study patients are evaluated at Weeks 0, 1, 2, 4, 8, 12 to Week 48 after being treated on one of the following regimens:

Stavudine (d4T) + Didanosine (ddI) + Lamivudine (3TC) or d4T + ddI + Indinavir or d4T + ddI + Nevirapine.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* Diagnosed asymptomatic HIV infection.
* HIV-1 RNA greater than 500 copies/ml.
* CD4+ T-cell count greater than 200/mm3.
* Never received antiretroviral therapy.

Exclusion Criteria

Co-existing Condition:

Excluded:

Severe non-HIV-related disease.

Patients with the following prior conditions are excluded:

History of neuropathy.

Prior Medication:

Excluded:

* Investigational drug within 1 month prior to study.
* Immunomodulatory drug within 1 month prior to study.

Prior Treatment:

Excluded:

* Radiation therapy within past month.
* Chemotherapy within past month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Cornell AIDS Clinical Trials Unit, New York, New York, United States

REFERENCES:
- [Background] Katlama C, Murphy R, Johnson V, Squires K, Horban A, Gatell J, Clotet B, Staszewski S, VanLeeuwen R, Clumeck N, Moroni M, Pavia A, Schmidt Au Gonzalez-Lahoz J, Antunes F, Gulick R, Banhegyi D, Montaner J, Calvez V, Sommadossi JP, Lange J. The Atlantic study: a randomised open-label study comparing two protease inhibitors (PI)-sparing antiretroviral strategies versus a standard PI-containing regimen. Conf Retroviruses Opportunistic Infect. 1999 Jan 31-Feb 4;6th:70 (abstract no 18)
- [Background] Norton M. Choosing the right initial antiretroviral regimens. GMHC Treat Issues. 1999 Feb;13(2):7-10. PMID 11366117
- [Background] Douglas J. Ward, MD. Lipodystrophy Substudy of Atlantic Trial Offers Limited Insights. http://www.medscape.com/viewarticle/438301
- [Background] Murphy RL, Katlama C, Weverling GJ, et al. Fat redistribution and metabolic changes with a nucleoside-reverse transcriptase inhibitor (NRTI), non-NRTI, or protease inhibitor-based regimen: FRAMS substudy of the Atlantic study. Program and abstracts of the XIV International AIDS Conference; July 7-12, 2002; Barcelona, Spain. Abstract WeOrB1306.